CLINICAL TRIAL: NCT06425523
Title: Strengthening Resilience to Climate Change by Improving Mental Health: Evidence from a Randomized Intervention in Southwestern Uganda
Brief Title: Transforming Health and Resilience in Vulnerable Environments: Mental Health, Psychosocial Support, and Climate-Smart Farming in Nakivale
Acronym: THRIVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Vivo international e.V. (Industry); Bielefeld University (Other); Kabale University (Other); University of Turku (Other); Max Planck Institute for Research on Collective Goods (Unknown); University of North Carolina, Charlotte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAK-SH/HGI-2024; 2022-01573_Formas (Other Grant/Funding Number: Formas - a Swedish Research Council for Sustainable Development)
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Psychological Distress; Malnutrition, Child; Dietary Deficiency; Mental Health; Malnutrition
Keywords: Self-Help Plus; Home Gardening Intervention; Uganda; Refugee; Nakivale; Mental health; Child development; Food security; Climate change adaptation; Climate smart agriculture; Farming intervention
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Three-arm, parallel-group, 1:1:1 allocation, superiority, cluster-randomized controlled trial (cRCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EUC (Active Comparator): Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- HGI (Experimental): Home Gardening Intervention
  Interventions: Behavioral: Home Gardening Intervention (HGI); Behavioral: Enhanced Usual Care (EUC)
- SH+/HGI (Experimental): Self-Help Plus in combination with Home Gardening Intervention
  Interventions: Behavioral: Home Gardening Intervention (HGI); Behavioral: Self-Help Plus (SH+); Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Home Gardening Intervention (HGI) — The Home Gardening Intervention (HGI) provides refugee participants with agricultural inputs and training (field prep., sowing, water management, pest control, weeding, etc.) through a participatory field school approach with a curriculum derived from best practices in agro-ecology. The program includes active monitoring during a 12-month period. The training involves nutrition education on cooking methods and the importance of dietary diversity using garden produce as well as guidance on surplus management and market support. The overall goal of the intervention is to enable climate-resilient farming for improved food security and dietary diversity that is sustainable long-term.
  Arms: HGI; SH+/HGI
Behavioral: Self-Help Plus (SH+) — Self-Help Plus (SH+) is a 5-session group intervention developed by the WHO and based on Acceptance and Commitment Therapy, delivered by trained local facilitators. It provides tools to manage stress and adversity through pre-recorded audio lessons and a self-help book. Sessions include individual exercises and group discussions.
  SH+ aims to decrease psychological distress. It has shown effectiveness among refugees in Uganda and elsewhere.
  Arms: SH+/HGI
Behavioral: Enhanced Usual Care (EUC) — The Enhanced Usual Care (EUC) control condition involves a single 15-minute psychoeducation session providing information on managing overthinking and utilizing available mental health services in the settlement. These services include psychosocial support from community health workers and clinical mental health services (counseling and medications) provided weekly at local primary care centers by a visiting team.

SUMMARY:
The study aims to evaluate if enhancing the mental health of refugee mothers can make them better able to implement new farming methods that are meant to improve food security in the face of climate change. It is a cluster-randomized controlled trial involving 900 pairs consisting of refugee mothers and their children aged 36-59 months, living in Nakivale refugee settlement in Uganda. The mothers will be randomly assigned to one of three groups:

* Control group: Mothers will receive Enhanced Usual Care (EUC).
* HGI group: Mothers will receive the Home Gardening Intervention, consisting of training and supplies for home gardening.
* HGI/SH+ group: Mothers will receive both the Home Gardening Intervention and the Self-Help Plus mental health intervention.

The main goal is to see if the gardening program alone can reduce food insecurity after 12 months compared to the EUC control group. It also aims to see if reducing psychological distress by adding the mental health component boosts the effects of the gardening intervention.

Secondary goals are to look at impacts on dietary diversity, child malnutrition, and mothers' mental health levels across all three groups.

The study also gathers survey data on participant mothers' migration history, social capital, exposure to potentially traumatic events, exposure to natural hazards and environmental stressors, mental health, and parenting style. Both mothers and their children will furthermore play incentivized economic games to measure their economic preferences (time, risk, social preferences). Additionally, the study will assess children's well-being and functioning. Children will also be asked to carry out gamified tasks designed to measure their cognitive development.

ELIGIBILITY:
Inclusion Criteria (mothers):

* Psychological distress (score 5 or above on K-6)
* Ability to speak and understand Kiswahili
* Have a child aged 36-59 months
* Availability of plot of land for farming
* Access of water for farming
* Written informed consent to enter the study

Exclusion Criteria (mothers):

* Imminent risk of suicide
* Observable signs of psychosis
* Manic behaviors
* Intellectual disability

Inclusion criteria (children):

* Age 36-59 months
* Written parental consent to enter the study
* Assent to enter the study

Exclusion criteria (children):

* Intellectual disability
* Not living with mother

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Food insecurity | 12 months
  Food insecurity will be assessed using the Food Insecurity Experience Scale (FIES). The FIES was developed by the FAO, and consists of 8 questions regarding the availability of sufficient food in the past thirty days. The questions form a scale calibrated against a global reference from the 2014-2016 Gallup World Poll for comparability across countries. Responses are analyzed as a scale using Item Response Theory (IRT) models, ensuring comparability of food insecurity prevalence rates.

SECONDARY OUTCOMES:
Dietary diversity | 12 months
  Dietary diversity will be assessed using the Household Dietary Diversity Score (HDDS). The HDDS is a measure of food consumption that reflects a household's access to a variety of foods. It's based on households' self-reporting of the 12 food groups consumed in the previous 24 hours.
Child malnutrition | 12 months
  Child malnutrition will be assessed using the Height-for-Age Z-score (HAZ). The HAZ is a standard statistical measurement that represents how a child's height compares to a reference population of the same age and sex. It's used to assess long-term nutritional status and can indicate chronic malnutrition or stunting. A HAZ score below -2 is considered stunted, indicating that the child is significantly shorter than the average height for their age. A score above +2 would suggest the child is taller than the average height for their age.
Psychological distress | 12 months
  Psychological distress will be measured using the Kessler Psychological Distress Scale (K6). The K6 is a concise tool used to screen for psychological distress. It assesses general psychological distress through six questions that inquire about symptoms of depression and anxiety experienced in the past month. Each of the six questions is scored from 0 (none of the time) to 4 (all of the time), providing a total score range from 0 to 24. Higher scores indicate greater psychological distress.

OTHER OUTCOMES:
Economic preferences | 12 months
  Both mothers and their children will play a set of incentivized economic games to measure economic preferences. Risk-taking will be measured using a "bomb-task." Time preferences will be measured using an investment task. Prosociality will be assessed using a series of dictator games.
Cognitive skills | 12 months
  Children's cognitive skills will be assessed using a battery of gamified tasks. Spatial cognition will be measured using 3d blocks and 2d shapes. Mathematics ability will be assessed using free counting, give-n, number comparison, and addition/subtraction tasks. Theory of mind will be measured using surprise content and surprise outcome tasks. Gaze following will be measured using TANGO. Language skills will be assessed using TIFALDI.
Social capital | 12 months
  Social capital will be measured using survey items asking about group membership, involvement in citizenship activities, and trust.
Positive parenting | 12 months
  Positive parenting will be assessed using the 6-item Positive Parenting Subscale of the Alabama Parenting Questionnaire (APQ). This subscale focuses on the frequency of positive interactions between parents and children. Each item is rated on a scale from 1 (never) to 5 (always), with higher scores indicating more frequent use of positive parenting practices.
Maltreatment | 12 months
  Child maltreatment will be measured using the 11-Item Discipline Module of the Multiple Indicator Cluster Survey (MICS). MICS is a household survey developed by UNICEF. It consists of eleven Yes/No questions that inquire about the different disciplinary actions taken by the caregiver in the past month. The total score can range from 0 to 11, with higher scores indicating the use of more types of disciplinary actions.
Posttraumatic stress | 12 months
  Posttraumatic stress will be measured using the Post-Traumatic Checklist 6-item Civilian Version (PCL-C). It has 6 items rated from 1 to 5, measuring key PTSD symptoms. Total score ranges from 6 to 30, with scores above 14 indicating potential PTSD.
Stress | 12 months
  Stress will be assessed with the Perceived Stress Scale 4-item version (PSS-4). The PSS-4 is a brief self-report measure of perceived stress. It consists of four questions that ask about feelings and thoughts during the last month. Each item is rated on a scale from 0 (Never) to 4 (Very often), with items 2 and 3 reverse scored. The total score, ranging from 0 to 16, is obtained by adding the scores of all items. Higher scores indicate higher perceived stress.
Depression | 12 months
  Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a widely-utilized questionnaire that gauges the severity of depression in individuals. It consists of nine items, each corresponding to a symptom of depression. The responses are scored on a scale ranging from 0 (not at all) to 3 (nearly every day), with the total score indicating the depression level. The scale's range is 0-27, reflecting varying degrees of depression severity from mild to severe.
Anxiety | 12 months
  Anxiety will be assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7). The GAD-7 is a brief measure designed to assess the severity of generalized anxiety disorder symptoms. It includes seven items that evaluate key symptoms such as nervousness, excessive worry, and fear. Respondents rate how often they have been bothered by each symptom over the past two weeks on a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 21, with higher scores indicating more severe anxiety.
Psychological flexibility | 12 months
  Psychological flexibility will be measured using the Acceptance and Action Questionnaire - version 2 (AAQ-2). The AAQ-2 consists of seven items scored on a 7-point Likert scale ranging from 1 (never true) to 7 (always true). The total score can range from 7 to 49, with higher scores indicating greater psychological inflexibility.
Functional impairment | 12 months
  Functional impairment will be assessed using a 15-item version of the World Health Organization Disability Assessment Schedule 2.0 (WHODAS-II). The WHODAS-II is a standardized instrument for measuring health and disability across various domains of functioning. It covers six domains: cognition, mobility, self-care, getting along, life activities, and participation. Each item is rated for difficulty over the past 30 days on a 5-point scale from 0 (none) to 4 (extreme or cannot do). The scores can be summed to provide a profile of functioning and disability.
Subjective wellbeing | 12 months
  Subjective wellbeing will be measured using the WHO-5 Well-Being Index. the WHO-5 is a concise self-report tool that measures an individual's subjective well-being. It contains five questions that assess positive mood, vitality, and general interests. The responses are scored on a scale from 0 (at no time) to 5 (all of the time), and the total score is then multiplied by 4 to give a final score ranging from 0 to 100. A score of 0 indicates very poor well-being, while 100 represents excellent well-being.
Child wellbeing and functioning | 12 months
  Child wellbeing and functioning will be assessed using one of two versions of the Kiddy-KINDL questionnaire, depending on the child's age. For children aged 3 to 4 years, the parent version consists of 24 items that cover six subscales: physical well-being, psychological well-being, self-worth, family, friends, and functioning in everyday life (school or preschool/kindergarten). The items are scored on a 5-point Likert scale from 1 (never) to 5 (all the time), and a total score is calculated to reflect overall health-related quality of life. For children aged 4 years and above, there is a self-report version of the Kiddy-KINDL which contains 12 items. This version also uses a 5-point Likert scale for responses, and it similarly assesses various dimensions of a child's well-being.
Child emotional and behavioral problems | 12 months
  The PSC-17 (Pediatric Symptom Checklist-17) is a brief, 17-item parent-reported screening tool for identifying emotional and behavioral problems in children aged 4-17. It includes three subscales: Internalizing (5 items, anxiety/depression), Externalizing (7 items, conduct/aggression), and Attention (5 items, impulsivity/inattention), rated on a 3-point scale (0-2). Scores range from 0 to 34, with ≥15 suggesting possible psychosocial dysfunction, and subscale cutoffs at Internalizing (≥5), Externalizing (≥7), and Attention (≥7).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hall, PhD, Principal Investigator — Uppsala University
Locations (1):
- Kabale University, Kabale, Western Region, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tol WA, Leku MR, Lakin DP, Carswell K, Augustinavicius J, Adaku A, Au TM, Brown FL, Bryant RA, Garcia-Moreno C, Musci RJ, Ventevogel P, White RG, van Ommeren M. Guided self-help to reduce psychological distress in South Sudanese female refugees in Uganda: a cluster randomised trial. Lancet Glob Health. 2020 Feb;8(2):e254-e263. doi: 10.1016/S2214-109X(19)30504-2. PMID 31981556
- [Background] Al Daccache M, Abi Zeid B, Hojeij L, Baliki G, Bruck T, Ghattas H. Systematic review on the impacts of agricultural interventions on food security and nutrition in complex humanitarian emergency settings. BMC Nutr. 2024 Apr 19;10(1):60. doi: 10.1186/s40795-024-00864-8. PMID 38641632
- [Derived] Hall J, Ainamani HE, Vassiliou PTB, Doring S, Gredeback G, Peltonen K, Scharpf F, Sen U, Sutter M, Walsh JI, Hecker T. Combining mental health and climate-smart agricultural interventions to improve food security in humanitarian settings: study protocol for the THRIVE cluster-randomized controlled trial with mothers in Nakivale refugee settlement, Uganda. Trials. 2025 Sep 1;26(1):331. doi: 10.1186/s13063-025-09042-y. PMID 40890859